CLINICAL TRIAL: NCT02882932
Title: Comparative Evaluation of Intra-operative Peritoneal Lavage With Super Oxidized Solution and Normal Saline in Peritonitis Cases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DR RIKKI SINGAL, Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/MMIMSR/68/14
Record Dates: First submitted 2016-07-16; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Peritonitis
Keywords: peritonitis; solutions; normal saline; infection; peritoneal lavage
MeSH Terms: conditions — Peritonitis; Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Super Oxidized Solution (Other): Procedure/Surgery: Super Oxidized Solution(SOS) in group I - SOS with normal saline solution was used
  Interventions: Procedure: Super Oxidized Solution in group I
- normal saline (Other): Procedure/Surgery: normal saline
  In group II - patients underwent normal saline wash and bacterial load was noted.
  Interventions: Procedure: Super Oxidized Solution in group I

INTERVENTIONS:
Procedure: Super Oxidized Solution in group I — Two groups were made as group I and group II. Peritoneal Lavage was given with SOS and normal saline in group I. in group II only normal saline wash was given.
  Other Names: normal saline solution

SUMMARY:
Super Oxidized Solution (SOS) was used in peritonitis and results were compared by using normal saline solution in two groups. Abdominal fluid was taken to check for bacterial load after giving lavage with SOS solution and in other group normal saline. SOS is a high level disinfectant, non-flammable and no special training is required to handle it.

DETAILED DESCRIPTION:
Aim - To investigate the efficacy of super-oxidized solution (SOS) over normal saline in peritonitis. The investigators objectives are to present the potential clinical impact of intraperitoneal lavage with solutions for early recovery of the patient by reducing the infection rate.

Methods - A double-blind random clinical trial was performed in 240 patients diagnosed as peritonitis at MMIMSR, Mullana, Ambala, India, from December 2014 - November 2015. Subjects were divided into 2 groups, i.e. 120 patients in the study group and 120 cases in the control group. Both the groups underwent peritoneal lavage ; the study group received SOS where as control group underwent normal saline lavage. The effectiveness of both the solutions were compared.

ELIGIBILITY:
Inclusion criteria:

* gastric, duodenal, ileal perforation, appendicitis
* those patients were willing to participate and the informed consent was taken

Exclusion criteria:

* evidence of enteric encephalopathy
* liver diseases
* renal diseases
* heart disease
* known allergy to any substance
* multiple trauma or organ injury
* any gynaecological etiology

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
the investigators measured the infection rate by checking the bacterial load during after surgery | average of one year
  The investigators asked about the infection, early recovery

SECONDARY OUTCOMES:
The Results Were Measured In the Form of the, Early Recovery, Early Bowel Sounds | With in 10 -20 days
  the condition of the patient measured in the form of early bowel sounds, fever and discharge from the operated area

IPD SHARING:
Plan to Share IPD: No